CLINICAL TRIAL: NCT05421390
Title: Effect of Dairy Products on Insulin Resistance in Overweight and Obese Individuals with Prediabetes
Brief Title: Effect of Dairy Products on Insulin Resistance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Dairy Farmers of Canada (Other)
Responsible Party: Principal Investigator, Sergio Burgos, Associate Professor, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-7468
Record Dates: First submitted 2022-06-13; First posted 2022-06-16 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Insulin Sensitivity; Glucose Intolerance; PreDiabetes
MeSH Terms: conditions — Insulin Resistance; Glucose Intolerance; Prediabetic State

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- ≤1 dairy serving/day (No Intervention): Limited dairy intake
- 2-3 servings/day reduced-fat (Experimental): 2-3 servings/day of skim milk, fat-free yogurt, and low-fat cheese
  Interventions: Other: Reduced fat dairy
- 2-3 servings/day regular-fat (Experimental): 2-3 servings/day of regular-fat milk, yogurt, and cheese
  Interventions: Other: Regular fat dairy

INTERVENTIONS:
Other: Reduced fat dairy — Serving sizes will be: 250 mL milk, 175 g yogurt, and 50 g cheese. Skim milk, fat-free yogurt, and ≤22 % fat cheese
  Arms: 2-3 servings/day reduced-fat
Other: Regular fat dairy — Serving sizes will be: 250 mL milk, 175 g yogurt, and 50 g cheese. 3.25% fat milk, ≥2% fat yogurt, and ≥28% fat cheese
  Arms: 2-3 servings/day regular-fat

SUMMARY:
The objective of the study is to determine the effect of dairy consumption on insulin sensitivity in overweight and obese adults with prediabetes. Men and women (30-65 y) will be recruited from the greater Montreal area. Upon screening, those with prediabetes will complete a 2-wk run-in period in which participants will consume 1 serving/d of reduced-fat dairy. Adherent participants will be randomized by sex into 1 of 3 groups: ≤1 serving/d of dairy (limited dairy) or 2-3 servings/d of reduced-fat or regular-fat dairy for 12 weeks. Participants will be instructed on how to incorporate foods into their diet in a manner that prevents changes in their body weight. The hyperinsulinemic-euglycemic clamp will be used before and after the intervention to document potential changes in insulin sensitivity as the primary outcome. In addition, glycemic variables, body composition, and cardiometabolic risk factors will be assessed as secondary outcomes. Serum lipidomic and global gene expression responses to the intervention in subcutaneous adipose tissue will be measured as exploratory variables. Adherence to intervention will be assessed at each visit by food diaries, a record of consumed dairy products, and serum proportion of 15:0, 17:0, and t16:1n7 fatty acids as objective biomarkers of dairy fat intake.

DETAILED DESCRIPTION:
The randomized controlled trial will be preceded by a 2-week run-in period in which participants will consume 1 serving/day of reduced-fat dairy. Following the run-in period, adherent participants will be randomly assigned to one of the three treatment groups (n=20 per group) in a 1:1:1 allocation ratio. Stratified permuted block randomization will be used to ensure adequate balance among groups using a computer-generated list of random numbers. Due to the nature of the test products, participants cannot be blinded to the diet intervention. However, outcome assessors will be blinded to treatment allocation.

During the screening visit, and after obtaining informed consent, eight, height, waist circumference, blood pressure, and pulse will be measured. Standard blood and urine tests, an OGTT, chest X-ray, electrocardiogram, and a physical exam will be performed. In addition, volunteers will be interviewed regarding demographic information, medical and family history, dietary habits, and physical activity using questionnaires.

At the run-in visit, participants will retrieve their dairy products and a dietitian will instruct them on how to incorporate incorporating 1 serving of reduced-fat dairy products each day into their habitual diet. Participants will be asked to record their food intake for 3 consecutive days (including one weekend day). They will also receive an accelerometer and instructions for use on the same 3-days they record their food intake. Participants will maintain a daily record of consumed dairy products during the run-in periods and throughout the study.

At the baseline and 12-week intervention visits, participants will undergo a hyperinsulinemic-euglycemic clamp to assess systemic insulin sensitivity. In addition, body composition will be measured by dual-energy X-ray absorptiometry and resting energy expenditure by indirect calorimetry. A biopsy of subcutaneous adipose tissue from the thigh will be taken at fasting.

During the 12-week intervention, participants in the limited dairy group will be instructed to limit their intake of dairy products to ≤1 serving/d of dairy. Participants in the 2-3 dairy servings of reduced or regular fat dairy groups will be provided with the study products. Serving sizes will be 250 mL milk, 175 g yogurt, and 50 g cheese. The dietitian will instruct participants individually on how to incorporate the dairy products into their habitual diets by reducing the intake of other foods of equivalent caloric content and complementary nutrient density, to maintain stable body weight. No additional dietary changes will be recommended.

At the monthly follow-up visits, weight, blood pressure, and pulse will be measured. In addition, participants will complete questionnaires about their health and physical activity. At each visit, they will be asked to track their food intake for 3 consecutive days (including one weekend day) using a mobile application on their smartphone or, if not possible, in written food diaries. Additionally, a blood sample will be collected to measure fatty acid biomarkers of dairy intake. On the second monthly visit, they will also receive an accelerometer and instructions for use on the same 3-days they record their food intake for the 12-week visit.

At the final follow-up visit, participants' weight, blood pressure, and pulse will be measured, and they will complete questionnaires regarding their health and activity. They will undergo an oral glucose tolerance test, as well as blood and urine tests, as described for the first visit.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 30 and 65 years,
* Able to provide informed consent,
* Stable weight and dietary habits over a period of 3 months,
* Body mass index of 25-40 kg/m2,
* Waist circumference ≥94 cm for men, ≥80 cm for women,
* One or more indicators of prediabetes:

  1. 5.7-6.4% HbA1c
  2. fasting 5.6-6.9 mmol/L glucose, or
  3. 7.8-11.0 mmol/L glucose at 2-h OGTT

Exclusion Criteria:

* Current smokers,
* Pregnant or planning to become pregnant in the next 6 months,
* Breastfeeding,
* Participation in a weight loss program in the past 3 months,
* Dairy allergy or lactose intolerance,
* Any diagnosed eating disorders,
* Substance abuse (drugs or alcohol >3 drinks/day),
* Diagnosed medical conditions such as cardiovascular disease, anemia, kidney disease, liver disease and any cancer, other than skin, within 5 years.
* Diabetes diagnosis,
* Abnormal electrocardiogram or chest X-Ray,
* Treatment with diuretics, certain β-blockers, bronchodilators, daily nonsteroidal anti-inflammatory drugs, anticoagulants or antiplatelet agents (except prophylactic aspirin 81 mg/d), antianginals, antiarrhythmics, oral steroids, or other medications known to affect glucose metabolism,
* Refusal to temporarily stop taking supplements (vitamin D, calcium, multivitamins, herbal remedies),
* Serum creatinine > 120 µmol/L,
* Hemoglobin < 120 g/L,
* Liver function tests ≥ 2× upper limit,
* Positive viral serology,
* Inaccessible veins.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-06-10 (Actual); Primary Completion 2024-10-18 (Actual); Study Completion 2024-10-18 (Actual)

PRIMARY OUTCOMES:
Change in whole-body insulin sensitivity | Difference between baseline and 12-weeks intervention visit
  Change in whole-body insulin sensitivity as measured by glucose infusion rate during the last 30 min of a hyperinsulinemic-euglycemic clamp divided by serum insulin concentration at the same period (M/I)

SECONDARY OUTCOMES:
Change in glucose tolerance | Difference between screening and 13-week follow-up visit
  Change in glucose tolerance as measured by plasma glucose concentration at 2-h oral glucose tolerance test
Change in Matsuda index | Difference between screening and 13-week follow-up visit
  Change in Matsuda index as measured by plasma glucose and insulin concentration during an oral glucose tolerance test
Change in Insulinogenic index | Difference between screening and 13-week follow-up visit
  Change in Insulinogenic index as measured by the ratio of serum c-peptide concentration and plasma glucose at 30 min minus 0 min during an oral glucose tolerance test
Change in oral disposition index | Difference between screening and 13-week follow-up visit
  Change in oral disposition index as measured by the product of the Matsuda index and Insulinogenic index
Change in Homeostatic Model Assessment for Insulin Resistance | Difference between screening and 13-week follow-up visit
  Change in Homeostatic Model Assessment for Insulin Resistance as calculated from fasting glucose and insulin concentration
Change in glycated hemoglobin | Difference between screening and 13-week follow-up visit
  Change in fasting serum glycated hemoglobin percent
Change in total lean body mass | Difference between baseline and 12-weeks intervention visit
  Change in total lean body mass as measured by dual-energy X-ray absorptiometry
Change in total fat mass | Difference between baseline and 12-weeks intervention visit
  Change in total fat mass as measured by dual-energy X-ray absorptiometry
Change in visceral fat mass | Difference between baseline and 12-weeks intervention visit
  Change in visceral fat mass as estimated by dual-energy X-ray absorptiometry
Change in systolic blood pressure | Difference between baseline and 12-weeks intervention visit
  Change in systolic blood pressure as measured by automated blood pressure monitor.
Change in diastolic blood pressure | Difference between baseline and 12-weeks intervention visit
  Change in diastolic blood pressure as measured by automated blood pressure monitor.
Change in total cholesterol | Difference between baseline and 12-weeks intervention visit
  Change in total cholesterol as measured by fasting serum concentration
Change in total triglycerides | Difference between baseline and 12-weeks intervention visit
  Change in total triglycerides as measured by fasting serum triglycerides
Change in total LDL-cholesterol | Difference between baseline and 12-weeks intervention visit
  Change in total LDL-cholesterol as measured as calculated from fasting serum total cholesterol, HDL-cholesterol, and triglycerides
Change in total HDL-cholesterol | Difference between baseline and 12-weeks intervention visit
  Change in total HDL-cholesterol as measured by fasting serum total HDL-cholesterol
Change in total non-HDL-cholesterol | Difference between baseline and 12-weeks intervention visit
  Change in total non-HDL-cholesterol as calculated from fasting serum total cholesterol and HDL-cholesterol
Change in C-reactive protein | Difference between baseline and 12-weeks intervention visit
  Change in fasting serum C-reactive protein concentration

OTHER OUTCOMES:
Change in resting energy expenditure | Difference between baseline and 12-weeks intervention visit
  Change in resting energy expenditure as measured by indirect calorimetry
Change in metabolic flexibility | Difference between baseline and 12-weeks intervention visit
  Change in metabolic flexibility as measured by the difference in respiratory quotient between basal and hyperinsulinemic periods of a hyperinsulinemic-euglycemic clamp
Change in total energy expenditure | Difference between baseline and 12-weeks intervention visit
  Change in total energy expenditure as measured by accelerometry
Change in metabolic equivalent of task | Difference between baseline and 12-weeks intervention visit
  Change in metabolic equivalent of task as measured by accelerometry
Change in total energy intake | Difference between baseline and 12-weeks intervention visit
  Change in total energy intake as calculated from 3-d food records
Change in dairy fat intake biomarkers | Difference between baseline and 12-weeks intervention visit
  Change in the proportion of 15:0, 17:0 and/or t16:1n7 fatty acids in serum lipid fractions
Change in serum lipidomic signatures | Difference between baseline and 12-weeks intervention visit
  Change in the concentration of serum lipid species as measured by liquid-chromatography mass spectrometry
Change in subcutaneous adipose tissue gene expression signature | Difference between baseline and 12-weeks intervention visit
  Change in the expression of genes in subcutaneous adipose tissue as measured by RNA sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Sergio A Burgos, PhD, Principal Investigator — RI-MUHC
Locations (1):
- RI-MUHC, Montreal, Quebec, Canada